CLINICAL TRIAL: NCT05673382
Title: CrisisCope: Internet-based CBT Intervention for Distress Related to Life Crises.
Brief Title: CrisisCope: ICBT for Psychological Symptoms Related to Life Crises.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Gerhard Andersson, Professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CrisisCope
Record Dates: First submitted 2023-01-04; First posted 2023-01-06 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-04

CONDITIONS: Depressive Symptoms; Anxiety Symptoms
Keywords: Life crises; Randomized controlled trial; Internet-based cognitive behavioral therapy (ICBT); Internet intervention; Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: After recruitment finished, participants will be randomized to either intervention condition (treatment group) or control condition (wait-list). Participants in the control condition will receive the same treatment once the treatment group has finished the treatment and outcome measures has been collected from both groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Eight weeks of individually tailored ICBT, were participants receives in total 8 modules out of 20 possible depending on their current problems and described situation with weekly support by a therapist.
  Interventions: Behavioral: Internet-based cognitive behavioral therapy
- Control group (No Intervention): The control group is a wait-list control condition. Participants are instructed to wait. After the treatment group has finished their treatment and post-treatment measures has been collected, the control group receive the same treatment as the treatment group got.

INTERVENTIONS:
Behavioral: Internet-based cognitive behavioral therapy — The intervention (the treatment) within this study is based on cognitive behavioral therapy principles and adapted to target psychological symptoms related to life crises. The 20 modules that the intervention consists of include psycho-educational texts as well as examples and exercises.
  Arms: Treatment group

SUMMARY:
The aim with this study is to investigate the effects of internet-based cognitive behavioral therapy (ICBT) on psychological symptoms related to one or more life crises. The target group is adults (18 years or older) who have symptoms of depression, anxiety, stress, or other psychological distress related to one or more life crises. The ICBT consists of eight modules during eight weeks with weekly support by a therapist and the treatment group will be compared to a wait-list control condition. Participants will be recruited in Sweden with nationwide recruitment.

DETAILED DESCRIPTION:
The study is a randomized controlled trial about the effects of ICBT aiming to target psychological symptoms related to one or more life crises. Primary outcome measures are depressive symptoms (measured with Beck Depression inventory-II) and anxiety symptoms (measured with Generalized Anxiety Disorder-7). Other outcome measures used will for example be about adaptability, stress symptoms, sleep problems, post traumatic stress symptoms and quality of life.

Because the psychological impact of a life crisis can be diverse, between different people and between different kinds of crises, a transdiagnostic individually tailored treatment will be used that has been tested in several previous trials. This treatment has been adopted to target psychological symptoms related to life crises.

ELIGIBILITY:
Inclusion Criteria:

* Experience psychological symptoms related to one or more life crises.
* 18 years or older
* Adequate ability to speak, read and write Swedish
* Having access to the internet and a smartphone, computer or other device

Exclusion Criteria:

* Severe psychiatric or somatic issues that makes participation harder or impossible
* Ongoing addiction
* Acute suicidality
* Other ongoing psychological treatment
* Recent (within the past three months) changes in dose of psychotropic medication or planned change during the treatment weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-01-19 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2024-06-24 (Estimated)

PRIMARY OUTCOMES:
Beck Depression Inventory-II | Change between Baseline, end of treatment after eight weeks and follow-up at 12 months after treatment termination.
  Measure of depressive symptoms. Range for the total sum is between 0 and 63 with a higher score score indicating a higher level of depressive symptoms. Clinical ranges for minimal, mild, moderate and severe major depressive disorder are considered to be 0-13, 14-19, 20-28, and 29-63 respectively.
Generalized Anxiety Disorder-7 | Change between baseline, end of treatment after eight weeks and follow-up at 12 months after treatment termination.
  Measure of anxiety symptoms and worry. When summing the points of the seven first questions, the scores are interpreted as mild, moderate and severe anxiety symptoms at 5-10, 11-15, and above 15 respectively

SECONDARY OUTCOMES:
Brief Adjustment Scale-6 | Change between baseline, end of treatment after eight weeks and follow-up at 12 months after treatment termination. Also, every week during the treatment weeks.
  A measure of general psychological adjustment, consisting of six items. The items are on a seven-point response scale with higher scores indicating lower general psychological adjustment.
Patient Health Questionnaire-9 | Change between baseline, end of treatment after eight weeks and follow-up at 12 months after treatment termination.
  Measure of depressive symptoms. Possible range for the total sum is 0 to 27 (created by summing up the scores from each item) with a higher score indicating higher levels of depression. Clinical cut-offs for mild, moderate, moderately severe and severe major depressive disorder are considered to be 5, 10, 15 and 20 respectively.
Perceived Stress Scale-14 | Change between baseline, end of treatment after eight weeks and follow-up at 12 months after treatment termination.
  A questionnaire that aims to measure symptoms of stress. It contains of 14 items that are scored on a range between 0 (never) and 4 (very often). The total score range is between 0-56 and a higher score reflects higher levels of perceived stress.
Insomnia Severity Index | Change between baseline, end of treatment after eight weeks and follow-up at 12 months after treatment termination.
  Measure of insomnia severity and symptoms of disordered sleep. Norm score ranges include low likelihood of sleep problems (0-7 points), some sleep problems (8-14 points), moderate sleep problems (15-21 points), severe sleep problems (22-28 points).
Alcohol Use Disorder Identification Test | Change between baseline, end of treatment after eight weeks and follow-up at 12 months after treatment termination.
  A ten-item scoring tool to assess alcohol consumption, drinking behaviors, and alcohol-related problems. Scores are ranging from 0-40 with higher scores indicating a higher level of alcohol use.
Impact of Events Scale-Revised | Change between baseline, end of treatment after eight weeks and follow-up at 12 months after treatment termination.
  Assesses subjective distress caused by traumatic events.Items are rated on a five-point scale from 0 (not at all) to 4 (extremely). Total score range between 0-88, with a higher score indicating more severe distress caused by the traumatic events.
Brunnsviken Brief Quality of Life Scale | Change between baseline, end of treatment after eight weeks and follow-up at 12 months after treatment termination.
  Measure of quality of life with a total score ranging from 0 to 96 with a higher score indicating higher quality of life. The scores of each of the six primary questions regarding perceived quality of life within an area of life are multiplied with the score of an item measuring the perceived importance of the area in question.
InCharge Financial Distress/Financial Well-Being Scale | Change between baseline, end of treatment after eight weeks and follow-up at 12 months after treatment termination.
  A measure aiming to measure distress related to the individual's economic situation. It consists of eight questions where the respondent gets to answer on a scale from 1 to 10.
Medical Outcome Study Social Support Survey | Change between baseline, end of treatment after eight weeks and follow-up at 12 months after treatment termination.
  A 12-item questionnaire aiming to measure the individual's perceived social support that is answered on a five-point scale (1-5). Besides the 12 items, the questionnaire also includes a question about how many family members and friends that the individual experience to have, who he/she can talk to. Total score range between 12 to 60.
Posttraumatic Growths Inventory-Short form | Change between baseline, end of treatment after eight weeks and follow-up at 12 months after treatment termination.
  A questionnaire consisting of 10 items, aiming to investigate the individual's experience of positive change in relation to challenging life events. Each item are answered on a six-point scale ranging between 0 to 5, resulting in a total score range between 0-60.

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Andersson, PhD, Principal Investigator — University Hospital, Linkoeping
Locations (1):
- Department of Behavioral Sciences and Learning, Linköping University, Linköping, Östergötland County, Sweden